CLINICAL TRIAL: NCT02283580
Title: Intramuscular and Functional Effects and Mechanism of Partitioning the Exercising Muscle Mass in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Low Load, High-repetitive Elastic Band Resistance Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Saey, Didier, M.D. (Individual); Maltais, Francois, M.D. (Industry)
Responsible Party: Principal Investigator, Andre Nyberg, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLHR-COPD-2014
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Healthy
Keywords: COPD; Healthy adults; Resistance training; Elastic bands; Limb muscle function; Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single limb resistance training (Experimental): Low load, high-repetitive resistance training.
  * single limb at a time (e.g., one arm or one leg)
  * elastic bands
  Interventions: Other: Single limb
- Two limb resistance training (Active Comparator): Low load, high-repetitive resistance training.
  * two limbs at a time (e.g., both arms or both legs)
  * elastic bands
  Interventions: Other: Two limb

INTERVENTIONS:
Other: Single limb — Low load, high-repetitive resistance training.
  * single limb at a time (e.g., one arm or one leg)
  * elastic bands
  * 8 weeks
  * 3 times/week,
  * each session 60 minutes
  * seven resistance exercises: Latissimus row, leg curl, elbow flexion, chestpress, plantar flexion, shoulder flexion and knee extension
  * maximal number of repetitions (RM) * 3 sets in each exercise.
  Arms: Single limb resistance training
Other: Two limb — Low load, high-repetitive resistance training.
  * two limbs at a time (e.g., both arms or both legs)
  * elastic bands
  * 8 weeks
  * 3 times/week,
  * each session 60 minutes
  * seven resistance exercises: Latissimus row, leg curl, elbow flexion, chestpress, plantar flexion, shoulder flexion and knee extension
  * maximal number of repetitions (RM) * 3 sets in each exercise.
  Arms: Two limb resistance training

SUMMARY:
Recent work have shown that low load, high-repetitive single limb resistance training, if compared to a control, can increase limb muscle function and functional exercise capacity in patients with chronic obstructive pulmonary disease (COPD) while avoiding the occurrence of limiting exertional symptoms. However, no comparison to another exercise regimen have been performed. In addition neither the intramuscular nor the mechanism of this exercise regimen have been investigated and represents the aim of the proposed project. We will in a prospective, assessor-blind; block randomized controlled, parallel-group trial compare single-limb to two-limb low load, high-repetitive resistance training in patients with severe and very severe COPD

The research hypothesizes are:

* that single-limb low-load high-repetitive resistance training will provide larger gain in the 6-min walking distance than two-limb low-load high- repetitive resistance training in patients with severe to very severe (stage III-IV) COPD.
* that eight weeks of single limb training should also be associated with larger physiological (increased muscle endurance, less muscle fatigue and deoxygenation) and structural (muscle protein synthesis, fiber-type distribution and capillarization) muscle adaptations to training, lower cardio- respiratory demand, as well a greater increase in health-related quality of life in comparison to two-limbs simultaneous training.

We will also compare the groups at baseline to investigate the acute effects and mechanisms of single-limb to two-limb low load, high-repetitive resistance training, a comparison that also will include healthy matched controls.

The research hypothesizes are:

* that involving a large muscle mass during exercise (e.g., two-limb low load, high-repetition resistance training) compared to involving a small muscle mass during training (e.g., single limb low load, high-repetition resistance training) would lead to larger restraints on the cardiorespiratory system in patients with severe to very severe COPD. Conversely, single limb interventions should produce less dyspnea and more muscle deoxygenation and fatigue than two-limb simultaneous exercise while healthy controls will be able to perform both legs/arms exercise without a central constraint, and no negative consequences on muscle fatigue or exercise stimulus.

ELIGIBILITY:
Inclusion criteria (COPD):

* Age: > 40
* Cumulative (current or ex) smoking history >10 pack-years
* COPD with non-reversible airflow obstruction corresponding to GOLD 3 and 4

Exclusion Criteria:

* Recent exacerbation (< 6 weeks)
* Neuromuscular and/or orthopedic disorders that compromises participation to an exercise program
* Recent cancer
* Unstable cardiac disease and cardiac stimulator
* Asthma
* Low body weight or obesity (Body Mass Index < 20 Kg/m2 and or > 30kg/m2)
* Significant hypoxemia at rest (SaO2 <85%)
* a daily dose > 10mg of systemic prednisone.

Inclusion criteria (Healthy controls)

* Age: > 40
* Normal pulmonary function tests.

Exclusion criteria

* Neuromuscular and/or orthopedic disorders that compromises participation to an exercise program
* Physically active (>9) according the Voorips questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Walking capacity (distance [meters]) | Baseline (week 0), 8 weeks
  Meters walked on the 6- minute walk test. The walking course will be 30 meters in length and the patients will be instructed in accordance to standardized guidelines to walk as far as possible in 6 minutes. One practice test will be performed to minimize risk of learning effect. The highest walking distance of the two 6-min walks will be chosen as baseline value.

SECONDARY OUTCOMES:
Unsupported upper extremity endurance capacity (time [seconds]) | Baseline (week 0), 8 weeks
  Endurance time (seconds) on the Unsupported Upper Limb Exercise test (UULEX) will be used to measure unsupported endurance capacity in the upper extremity. Participants will hold a plastic bar (0.2 kg), at shoulder width and will be asked to raise it from hip to the UULEX eight level chart for one minute at each level with a cadence of 30 movements per minute. If a patient reaches the highest level, the plastic bar will be replaced by a heavier one every minute. There are five different weights of the bar (0.2, 0.5, 1, 1.5, 2 Kg) and the patient will continue on the highest level until symptom limitation.
Isokinetic limb muscle function (Endurance [total work], strength [peak torque]) | Baseline (week 0), 8 weeks
  Isokinetic limb muscle function during one-arm shoulder flexion, one-leg knee extension and two-leg knee extension will be assessed. The subjects are informed to flex their arm or extend their leg(s) 25 consecutive times using maximal effort at each repetition during the concentric phase and to rest during the eccentric phase of the movement. Two different aspects of isokinetic muscle function will be measured. Peak torque from the highest contraction will be used for maximal strength and the total work generated from all contractions will be used for limb muscle endurance. The tests will be performed at an angular velocity of 60°• s-1,
Ventilatory response | Baseline (week 0), 8 weeks
  Respiratory response during all elastic band exercises (1: one-arm shoulder flexion, biceps flexion, chest press and latissimus row 2: two-arm shoulder flexion, biceps flexion, chest press and latissimus row 3: one-leg knee extension, plantar flexion and leg curl 4: two-leg knee extension, plantar flexion and leg curl) will be determined using a portable gas analysis system (Oxycon Mobile, Viasys Healthcare, Jaeger, Germany. Minute ventilation (VE) oxygen uptake (VO2), carbon dioxide excretion (VCO2,), heart rate (HR), respiratory exchange ratio (RER) and pulsed oxygen saturation (SpO2) will be collected
Cardiac output | Week 0 and week 8
  Arterial blood pressures and cardiac output will be non-invasively measured by a finger photoplethysmography device (BMEYE, Nexfin HD, Academic Medical Center, Amsterdam, The Netherlands) during all elastic band exercises detailed above.
Muscle deoxygenation | Baseline (week 0), week 8
  Changes of deoxyhemoglobin/myoglobin concentrations will be non-invasively measured by near-infrared spectroscopy of vastus lateralis muscle. Obtained during all elastic band exercises detailed above
Dyspnea (Rating [0-10]) | Baseline (week 0), 8 weeks
  Magnitude of dyspnea after each exercise and test will be measured by the Borg CR 10 scale
Limb muscle fatigue (Rating [0-10]) | Baseline (week 0), 8 weeks
  Magnitude of limb muscle fatigue after each exercise and test will be measured by the Borg CR 10 scale
Isometric muscle strength (maximum voluntary isometric contraction [MVIC], and supramaximal twitch tension (TW) and muscle fatigue | Baseline (week 0), 8 weeks
  Directly before and after all elastic band exercises (1: one-arm shoulder flexion, 2: two-arm shoulder flexion, 3: one-leg knee extension, 4: two-leg knee extension) generated force of both MVIC and TW will be measured by an isometric force gauge while participants will be in a standardized positioning. The occurrence of quadriceps (knee extension) or deltoid (shoulder flexion) fatigue induced by the exercise regimens will be quantified by measuring the fall in both MVIC and TW 15 after the elastic band resistance exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ); Didier Saey, Pht, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ)
Locations (2):
- Canada (2):
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Centre de recherche de l'IUCPQ, Québec

REFERENCES:
- [Derived] Nyberg A, Martin M, Saey D, Milad N, Patoine D, Morissette MC, Auger D, Stal P, Maltais F. Effects of Low-Load/High-Repetition Resistance Training on Exercise Capacity, Health Status, and Limb Muscle Adaptation in Patients With Severe COPD: A Randomized Controlled Trial. Chest. 2021 May;159(5):1821-1832. doi: 10.1016/j.chest.2020.12.005. Epub 2020 Dec 13. PMID 33316237
- [Derived] Nyberg A, Saey D, Martin M, Maltais F. Muscular and functional effects of partitioning exercising muscle mass in patients with chronic obstructive pulmonary disease - a study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:194. doi: 10.1186/s13063-015-0698-x. PMID 25927288